CLINICAL TRIAL: NCT07276776
Title: An Evaluation of the Omnipod® M System in Adults With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evolution 3
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; T2D; Omnipod 5; Automated Insulin Delivery System
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental- Participants with Type 2 diabetes (Experimental)
  Interventions: Device: Omnipod M system

INTERVENTIONS:
Device: Omnipod M system — The Omnipod M system will allow user to use a lower glucose target and improve systems glucose control

SUMMARY:
This is a single arm feasibility study to evaluate the Omnipod M System in adults with Type 2 Diabetes with the aim to enroll to 40 participants aged 18-75 years with type 2 diabetes to have a minimum of 20 participants initiate the use of Omnipod M System and the goal of 16 participants completing the 6-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18-75 years (inclusive)
2. Clinical diagnosis, based on investigator assessment, of type 2 diabetes for at least 6 months at time of screening
3. On current insulin regimen for at least 3 months prior to screening (i.e. basal-bolus, basal insulin only or premix)
4. Basal-bolus (AID or non-AID pump & MDI) or premix users with A1C < 14% OR basal users on long or intermediate acting insulin only with A1C > 8.0% and < 14%
5. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novolog, Admelog, Kirsty, Fiasp, Lyumjev or their generic equivalents
6. Deemed appropriate for pump therapy per Investigator's assessment considering previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
7. If using noninsulin glucose-lowering medications (such as GLP-1 receptor agonist, SGLT2 inhibitor, or other) or weight-reduction medications, dose has been stable for 6-weeks prior to screening; and participant is willing to not change the dose unless required for safety purposes.
8. Investigator has confidence that the participant can safely operate all study devices and can adhere to the protocol
9. Willing to wear the system, including Pods, continuously throughout the study
10. Willing and able to sign the Informed Consent Form (ICF)
11. Able to read and understand English
12. If of childbearing potential, willing and able to have pregnancy testing

Exclusion Criteria:

1. Any medical condition, which in the opinion of the Investigator, would put the participant at an unacceptable safety risk. This may include untreated malignancy, unstable cardiac disease, unstable or end-stage renal disease, unstable proliferative retinopathy, unstable psychiatric conditions such as eating disorders, drug or alcohol abuse.
2. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the 12 months prior to screening
3. Any planned surgery during the study which could be considered major in the opinion of the Investigator
4. History of more than 1 severe hypoglycemia in the past 6 months. Severe hypoglycemia is defined as an event that requires the assistance of another person due to altered consciousness, and requires another person to actively administer carbohydrate, glucagon, or other resuscitative actions
5. History of more than 1 diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS) in the past 6 months, unrelated to an intercurrent illness; kinked, dislodged, or occluded cannula; or initial diabetes diagnosis
6. Unable to tolerate adhesive tape or has any unresolved skin condition that could impact sensor or pump placement
7. Blood disorder or dyscrasia within 3 months prior to screening, which in the Investigator's opinion could interfere with determination of HbA1c
8. Use of hydroxyurea
9. Plans to receive blood transfusion over the course of the study
10. Pregnant or lactating, or is of childbearing potential and not using an acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilization such as tubal ligation or hysterectomy, or vasectomized partner); childbearing potential means that menstruation has started, and the participant is not surgically sterile or greater than 12 months post-menopausal).
11. Has taken systemic corticosteroids (oral or injectable) within 4 weeks or has had a local steroid injection (intraarticular, epidural) within 1 week prior to screening or plans to take oral or injectable steroids during the study
12. Participation in another clinical study using an investigational drug or device within 30-days or intends to participate in any other study during this study period
13. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the Investigator's clinical judgment
14. Participant is an employee of Insulet, an Investigator or a member of Investigator's study team, or immediate family member of any of the aforementioned

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Percent of time in hypoglycemic range <70mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Percent of time in hyperglycemic range >180 mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system

SECONDARY OUTCOMES:
Mean Glucose | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Percentage of time <54 mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Percentage of time >250mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Percentage of time >300mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Percent of time between 70-180mg/dL | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Standard Deviation | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the standard deviation (SD)
Coefficient of Variation | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV)
Average total daily insulin (TDI) | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Average TDI/kg | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system
Change in weight | Comparing baseline metrics to the end of the treatment period (Day45)
  measures change in weight
Patient reported outcomes | Comparing baseline metrics to the end of the treatment period (Day45)
  Participant responses to various questionnaires related to the investigational device as well as managing diabetes
4-hour post prandial glycemic metrics | Comparing baseline metrics to the end of the treatment period (Day45)
  Glucose metric from study continuous glucose monitoring system

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Joslin Diabetes, Boston, Massachusetts
  - MassResearch LLC., Waltham, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Mountain Area Health Educational Center ( MAHEC), Asheville, North Carolina
  - Texas Diabetes and Endocrinology (TDE), Austin, Texas
  - Disease & Glandular Disease Clinic, San Antonio, Texas